CLINICAL TRIAL: NCT05399069
Title: An Open-Label Safety Study of Single-dose VGR-R01 in Patients With Bietti Crystalline Dystrophy
Brief Title: Safety and Tolerability of VGR-R01 in Patients With Bietti Crystalline Dystrophy
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Tongren Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VGR-R01-001
Record Dates: First submitted 2022-05-11; First posted 2022-06-01 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-04

CONDITIONS: Bietti Crystalline Dystrophy
MeSH Terms: conditions — Bietti Crystalline Dystrophy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VGR-R01 (Experimental): Subretinal injection of VGR-R01
  Interventions: Drug: VGR-R01

INTERVENTIONS:
Drug: VGR-R01 — Gene Replacement Therapy

SUMMARY:
An Open-Label, Non-Randomized, Uncontrolled, Single-dose Pilot Study of VGR-R01 in Patients with Bietti Crystalline Dystrophy.

DETAILED DESCRIPTION:
VGR-R01 is a novel AAV vector carrying the human CYP4v2 coding sequence. This study is intended to evaluate the safety and tolerability of a single subretinal administration of VGR-R01. All subjects will undergo 365(±7) days of safety observation and will be encouraged to enroll in an extension study to evaluate the long-term safety of VGR-R01 for a total of five years.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years and <80 years of age;
2. Confirmed diagnosis of Bietti Crystalline Dystrophy;
3. Molecular diagnosis of CYP4v2 mutations (homozygotes or compound heterozygotes);
4. BCVA ≤ 20/200 in the study eye;
5. -8 D <diopters< +8 D, 21 mm < axial lengths ≤ 28 mm in the study eye;
6. Normal liver function and renal function；
7. Agree to use reliable barrier contraception for 1 year after administration of VGR-R01;
8. Able to provide informed consent and comply with requirements of the study. -

Exclusion Criteria:

1. Have insufficient viable retinal photoreceptor cells based on investigator's decision;
2. Have current ocular or periocular infections, or endophthalmitis;
3. Have any significant ocular disease/disorder other than BCD, including age-related macular degeneration, diabetic retinopathy, optic neuropathy, significant lens opacity, glaucoma, uveitis, retinal detachment, etc;
4. Have intraocular surgery history except cataract surgery in the study eye;
5. Prior medications which may interfere with the interpretation of study endpoints within six months before screening, eg. anti-VEGF drugs;
6. Have or potentially require of systemic medications that may cause eye injure;
7. Live attenuated vaccines is expected to be required during the study;
8. Participation in a clinical study with an investigational drug or medical device within three months before enrollment;
9. History of allergy or sensitivity to investigational drug, medications planned for use in the study;
10. Use of anticoagulants, or after 10 days cessation of anti-platelet agents the platelet function does not recover;
11. Use of any corticosteroids, other immunosuppressive drug(s) or antipsychotic drugs (eg. antidepressant, etc.) within 3 months prior to enrollment;
12. Have contraindications for corticosteroids or immunosuppressant;
13. Have complicating systemic diseases that would preclude the planned follow-up;
14. Abnormal coagulation function or other clinically significant abnormal laboratory results;
15. Have malignancies or history of malignancies;
16. History of immunodeficiency (acquired or congenital);
17. Females in lactation period;
18. Have a history of alcohol or illicit drug addiction;
19. Unable or unwilling to comply with the schedule of visits. -

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Estimated)
Dates: Start 2022-09-15 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Baseline up to Day 365
  An adverse event (AE) is any untoward medical occurrence in a clinical investigation participant administered a product; the event will not need to have a causal relationship with the treatment.
Incidence of serious adverse events | Baseline up to Day 365
  A serious adverse event (SAE) is any untoward medical occurrence at any dose that resulted in death; life threatening; require inpatient hospitalization or prolongation of existing hospitalization; result in persistent or significant disability/incapacity; result in congenital anomaly/birth defect.
Number of Participants with Clinically Significant Change from Baseline in Vital Signs | Baseline up to Day 365
  Vital signs (temperature, respiratory rate, pulse rate, systolic and diastolic blood pressure) will be obtained with participant in the seated position, after having sat calmly for at least 5 minutes. Clinical significance of vital signs will be determined at the investigator's discretion.
Number of Participants with Clinically Laboratory Abnormalities | Baseline up to Day 365
  Laboratory Tests will include hematology, coagulation, blood chemistry, urinalysis, serology, and pregnancy test, etc. If any potential changes accompanied by clinical symptoms, or results in a change of medical intervention, the findings will be considered as clinically significant based on investigator's decision.
Number of Participants with Clinically Significant Change from Baseline in Ophthalmic Examination Findings | Baseline up to Day 365
  Ophthalmic Examination will include BCVA, IOP, slitlamp examination, angiography and SD-OCT, etc. If any potential changes accompanied by clinical symptoms, or results in a change of medical intervention, the findings will be considered as clinically significant based on investigator's decision.

SECONDARY OUTCOMES:
Best-Corrected Visual Acuity (BCVA) | Up to Day 365
  BCVA will be assessed for both eyes using the Early Treatment of Diabetic Retinopathy Study (ETDRS) visual acuity (VA) chart. BCVA test should be performed prior to pupil dilation, and distance refraction should be carried out before BCVA is measured. Initially, letters are read at a distance of 4 meters from the chart. If <20 letters are read at 4 meters, testing at 1 meter should be performed. BCVA is to be reported as number of letters read correctly by the participant using the ETDRS Scale (ranging from 0 to 100 letters) in the study eye. The lower the number of letters read correctly on the eye chart, the worse the vision (or visual acuity). An increase in the number of letters read correctly means that vision has improved.
Changes from baseline in Visual Field indexes | Up to Day 365
  The outcome measeures will be assessed by Humphery perimetry
Changes from baseline in Microperimetry indexes | Up to Day 365
  The Microperimetry will be applied to assess the retinal sensitivity and the fixation behaviour.
Changes from baseline in ERG indexes | Up to Day 365
  The measeurement will be performed based on the standards of International Society for Clinical Electrophysiology of Vision (ISCEV)
Changes from baseline in m-ERG indexes | Up to Day 365
  The measeurement will be performed based on the standards of International Society for Clinical Electrophysiology of Vision (ISCEV)
Change from Baseline in NEI Visual Function Questionnaire (NEI-VFQ-25) | Up to Day 365
  NEI-VFQ-25 questionnaire measures dimensions of self-reported vision-targeted health status that are most important to persons with eye disease. Total score ranges from 0-100, where a score of 0 represents the worst outcome and 100 represents the best outcome.
Changes from Baseline in Spectral Domain Optical Coherence Tomography (SD-OCT) | Up to Day 365
Changes from Baseline in Optical Coherence Tomography Angiography(OCT-A) | Up to Day 365

CONTACTS AND LOCATIONS:
Overall Officials: Wenbin Wei, Principal Investigator — Vice President of Beijing Tongren Hospital
Locations (1):
- Beijing Tongren Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared with other researchers when VGR-R01 is fully approved.
Supporting Information: Study Protocol, SAP
Time Frame: IPD will be shared with other researchers when VGR-R01 is fully approved.
Access Criteria: IPD will be shared with other researchers when VGR-R01 is fully approved.